CLINICAL TRIAL: NCT05120804
Title: Improving Family Functioning in Obesity Treatment for Mexican American Women
Brief Title: Family Functioning in Obesity Treatment for Mexican Americans
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Becky Marquez (Other)
Responsible Party: Sponsor-Investigator, Becky Marquez, Assistant Professor, University of California, San Diego
Organization: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 210620
Record Dates: First submitted 2021-10-11; First posted 2021-11-15 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard behavioral treatment (Active Comparator): Nutrition and physical activity education along with behavior modification techniques
  Interventions: Behavioral: Standard behavioral treatment
- Standard behavioral treatment plus relationship skills training (Experimental): Nutrition and physical activity education along with behavior modification techniques plus brief and structured counseling on family functioning
  Interventions: Behavioral: Standard behavioral treatment plus relationship skills training

INTERVENTIONS:
Behavioral: Standard behavioral treatment — Nutrition and physical activity education along with behavior modification techniques
  Other Names: SBT
  Arms: Standard behavioral treatment
Behavioral: Standard behavioral treatment plus relationship skills training — Nutrition and physical activity education along with behavior modification techniques plus relationship skills training
  Other Names: SBTR
  Arms: Standard behavioral treatment plus relationship skills training

SUMMARY:
Mexican American families share similar elevated risks for obesity and obesity-related conditions, such as type 2 diabetes. Because negative family interactions and relationships (e.g., poor communication, high conflict, low emotional closeness) are associated with obesity treatment outcomes, this study tests a behavioral weight management intervention that provides relationship skills counseling to mothers and adult daughters. The goal is to improve family interaction patterns to buffer challenges and strengthen collaboration for eating and physical activity behaviors that support long-term weight management and thus provide an effective obesity treatment approach to address a major public health concern.

DETAILED DESCRIPTION:
Mexican American women are disproportionately affected by obesity and obesity-related conditions, such as type 2 diabetes. Obesity and diabetes are highly concordant in Mexican American families. Given the younger age of onset of diabetes in women with familial history, targeting mothers and their adult daughters for obesity treatment is warranted. From a family systems perspective, family-level approaches to obesity treatment can improve the adoption and maintenance of weight management behaviors. Including family members in treatment may also serve as a culturally salient intervention strategy as Mexican Americans endorse high level of familism. In contrast to traditional individual-level approaches to obesity treatment, a family-level approach grounded in familism would promote shared goals, collaborative problem solving, and communal coping when treating family members alongside each other. An important construct to consider when working with intergenerational Mexican American families is differences in acculturation, which may translate into differences in attitudes and behaviors. A wider gap in acculturation between parent and child has previously been associated with lower family functioning (e.g., poor communication, high conflict, low cohesion). However, interventions that promote bicultural competence by changing interactional patterns have been effective at improving family functioning. Hence, this study will conduct a randomized control trial testing the efficacy of a behavioral weight management intervention with brief and structured counseling on family functioning. Mexican American mothers and adult daughters (n=118 dyads) will be randomly assigned to receive standard behavioral treatment (SBT) or standard behavioral treatment plus relationship skills training (SBTR). Dyads participating in SBT or SBTR will attend 24 weekly sessions focused on nutrition and physical activity education along with behavior modification techniques. Dyads participating in SBTR will also receive experiential-based relationship skills training that draws from both general family systems concepts and behavioral family/couples therapy approaches to support familism, biculturalism, and communication competencies. The 12-month trial will consist of an intervention phase (1-6 months) and a maintenance phase (7-12 months). Assessments will be conducted at baseline and at the end of the intervention and maintenance phases. The primary outcome is weight loss. Secondary outcomes include treatment adherence (session attendance and self-monitoring records), physiological indicators of diabetes risk (hemoglobin A1c, waist circumference, and body fat percentage), health behaviors (eating and physical activity), psychological well-being (depression and perceived stress), and family functioning (subjective self-report and objective behavioral coding). Dyads in the SBTR group are expected to achieve greater improvements in primary and secondary outcomes than the STB group. Additionally, mediation by family functioning of intervention effects on primary and secondary outcomes will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-65 years of age
* Mexican or Mexican American
* Reside in San Diego County
* Body mass index of 25-45 kg/m2

Exclusion Criteria:

* Unable to read and write in English or Spanish
* Pregnant or plan to become pregnant in the next year
* Have a physical limitation that makes exercise like walking difficult
* Currently participating in a weight loss program
* Underwent weight loss surgery
* Report a serious medical or psychological condition

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identify as female
Enrollment: 236 (Estimated)
Dates: Start 2022-02-22 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Weight change | baseline to 6 month post-intervention
  Weight loss

SECONDARY OUTCOMES:
Weight change | 6 month post-intervention to 12 month follow-up
  Weight loss maintenance
Anthropometric measurement | baseline to 6 month post-intervention and 12 month follow-up
  Percent body fat
Hemoglobin A1C | baseline to 6 month post-intervention and 12 month follow-up
  Percent A1C
Family functioning | baseline to 6 month post-intervention and 12 month follow-up
  Observational coding of family communication
Eating behavior | baseline to 6 month post-intervention and 12 month follow-up
  Food frequency questionnaire
Physical activity | baseline to 6 month post-intervention and 12 month follow-up
  Accelerometer
Psychosocial factors | baseline to 6 month post-intervention and 12 month follow-up
  PHQ9

CONTACTS AND LOCATIONS:
Locations (1):
- University of California San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No